CLINICAL TRIAL: NCT05151653
Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Rising Intravenous Infusion or Subcutaneous Injection Doses of BI 765250 in Healthy Male Subjects (Single-blind, Randomised, Placebo-controlled, Parallel Group Design)
Brief Title: A Study to Test How Well Healthy Men Tolerate BI 765250 When Given as an Infusion Into the Vein or as an Injection Under the Skin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1474-0001; 2021-001727-40 (EudraCT Number)
Record Dates: First submitted 2021-12-01; First posted 2021-12-09 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BI 765250 arm (Experimental)
  Interventions: Drug: BI 765250
- Placebo arm (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 765250 — BI 765250
  Arms: BI 765250 arm
Drug: Placebo — Placebo
  Arms: Placebo arm

SUMMARY:
The main objectives of this trial are to investigate safety, tolerability, pharmacokinetics and pharmacodynamics following single rising doses of BI 765250.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 55 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the trial, in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetre of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders assessed as clinically relevant by the investigator
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections Further exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 139 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2024-09-13 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with treatment-emergent adverse events assessed as drug-related by the investigator | Up to 172 days

SECONDARY OUTCOMES:
Area under the concentration-time curve of the analyte in serum over the time interval from 0 extrapolated to infinity (AUC0-∞) | Up to 169 days
Maximum measured concentration of the analyte in serum (Cmax) | Up to 169 days

CONTACTS AND LOCATIONS:
Locations (1):
- SGS Life Science Services - Clinical Research, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com